CLINICAL TRIAL: NCT02286648
Title: Success Rate Evaluation of Miniature Pulpotomy With MTA in Primary Molars
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hossein Nematollahi, principal investigator, Mashhad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 921762
Record Dates: First submitted 2014-04-25; First posted 2014-11-10 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Pulpitis; Dental Pulp Disease; Tooth Diseases
Keywords: clinical signs; child; pulpotomy
MeSH Terms: conditions — Pulpitis; Dental Pulp Diseases; Tooth Diseases; Signs and Symptoms | interventions — formocresol; mineral trioxide aggregate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mineral Trioxide Aggregate (Experimental): pulpotomy with MTA
  Interventions: Drug: Mineral Trioxide Aggregate
- Formocresol (Active Comparator): pulpotomy with FC
  Interventions: Drug: Formocresol

INTERVENTIONS:
Drug: Formocresol — pulpotomy with formocresol
  Arms: Formocresol
Drug: Mineral Trioxide Aggregate — pulpotomy with MTA
  Arms: Mineral Trioxide Aggregate

SUMMARY:
The purpose of this study is to evaluate the clinical and radiographic success rate of Miniature pulpotomy with Mineral Trioxide Aggregate (MTA) in primary molars.

ELIGIBILITY:
Inclusion Criteria:

* healthy people(without any systemic disease)
* teeth :

  * no clinical or radiographic evidence of pulp degeneration
  * the possibility of proper restoration of the teeth

Exclusion Criteria:

* teeth :

  * excessive bleeding from the exposure site
  * internal root resorption
  * interradicular and/or periapical bone destruction
  * swelling or sinus tract

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
successful outcome of treatment as indicated by clinical signs defined with observation and check list | up to 12 months
  success or failure of treatment defined with observation and check list

SECONDARY OUTCOMES:
successful outcome of treatment as indicated by radiographic signs defined with observation and check list | up to 12 months
  success or failure of treatment defined with observation and check list

CONTACTS AND LOCATIONS:
Locations (1):
- Mashhad University of Medical Siences, Mashhad, Khorasan Razavi, Iran